CLINICAL TRIAL: NCT00729404
Title: Multicenter, Open-label, Randomized, Uncontrolled Study to Evaluate Inhibition of Ovulation of Two Transdermal Patch Formulations Containing 0.55 mg EE and Either 1.05 or 2.1 mg GSD in Healthy Young Female Vol. Over a Period of 3 Treatment Cycles
Brief Title: Inhibition of Ovulation, Patch, Ethinylestradiol and Gestodene
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91558; 2008-001198-13 (EudraCT Number)
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Contraception; Ovulation Inhibition
Keywords: Female Contraception; Ovulation Inhibition
MeSH Terms: interventions — Ethinyl Estradiol; Gestodene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestodene (BAY86-5016)
- Arm 2 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestodene (BAY86-5016)

INTERVENTIONS:
Drug: Ethinylestradiol/Gestodene (BAY86-5016) — transdermal patch: 0.55mg EE+2.1mg GSD; 3x7 days patch- wearing phase and a patch-free interval of 7 days (1 pre-treatment cycle, 3 treatment cycles)
  Arms: Arm 1
Drug: Ethinylestradiol/Gestodene (BAY86-5016) — transdermal patch: 0.55mg EE+1.05 mg GSD; 3x7 days patch- wearing phase and a patch-free interval of 7 days (1 pre-treatment cycle, 3 treatment cycles
  Arms: Arm 2

SUMMARY:
Investigation of two transdermal hormone patch formulations for contraception regarding inhibition of ovulation over a period of 3 treatment cycles in healthy young female volunteers

DETAILED DESCRIPTION:
Study was suspended due to inconclusive toxicology findings regarding the used patch formulation to be clarified prior to re-start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* BMI: 18 - 30 kg/m²,
* Healthy female volunteers,
* Age 18-35 years (smoker not older than 30 years, inclusive),
* Ovulatory pre-treatment cycle, at least 3 month since delivery,
* Abortion or lactation before the first screening examination,
* Willingness to use non-hormonal methods of contraception during entire study

Exclusion Criteria:

* Contraindications for use of combined (estrogen/gestodene) contraceptive (e.g. history of venous/arterial thromboembolic disease
* Regular intake of medication other than OCs
* Clinically relevant findings (blood pressure, physical and gynaecological examination, laboratory examination)
* Anovulatory pre-treatment cycle

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the proportion of volunteers with ovulation in at least one of the treatment cycles 2 and 3. | 4 month

SECONDARY OUTCOMES:
Assessment of ovarian activity during treatment cycle2 and 3 (Hoogland score) | 4 month
Course of gonadotropins (FSH, LH, P, E2) | 4 month
Endometrial thickness | 4 month
Follicle size | 4 month
Pharmacokinetics of EE, GSD and SHBG in treatment cycles 2 and 3 | 4 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/